CLINICAL TRIAL: NCT01762683
Title: Study of Role of Mononuclear Cells of Maternal Peripheric Blood in Human Myometrial Primar Cell Lines Differentiation Toward a Contratyl Phenotype: Influence of Preconceptional Obesity
Brief Title: Influence of Preconceptional Obesity on the Myometrial Cells Differentiation Toward a Contractyl Phenotype
Acronym: ObeDi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LIRUSSI-AOI-2011
Record Dates: First submitted 2012-05-31; First posted 2013-01-08 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pregnancy Complication
Keywords: pregnancy; obesity; differentiation
MeSH Terms: conditions — Pregnancy Complications; Obesity | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- pre-conceptional obesity with a scheduled cesarean section (Experimental)
  Interventions: Other: Myometrium biopsy and blood samples
- non-obese women with a scheduled cesarean section (Active Comparator)
  Interventions: Other: Myometrium biopsy and blood samples
- women entering labour (Active Comparator): women entering labour for vaginal delivery and for vaginal delivery
  Interventions: Other: Myometrium biopsy and blood samples

INTERVENTIONS:
Other: Myometrium biopsy and blood samples — The biopsy of myometrium is specially realised for the study in surgical unit after the release of the child, in women with normal pregnancy but necessitating a caesarean.
  The blood samples are realised, specially for the study, either during the medical exam before the ceasarean or specifically for the study.

SUMMARY:
The purpose of this study is to improve the understanding of cellular mecanism involved in delivery disorders in obese women, first by characterizing the hyperplasia phenomenon of myometrail cells induced by inflammatory stimulation (Il-1B), then by studying the role of blood mononuclear cells, of leptine and of obese women sera to interfere with the transition of myometrial cells toward hyperplasia phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed
* Patient affiliated with a social security scheme
* In front of for obstetrical reasons to give birth by caesarean section (scheduled caesarean section)
* Or a woman who is not obese in labour and needs to undergo a cesarean section
* No obvious infectious context
* Age > 18 years old

Exclusion Criteria:

* Obvious inflammatory or autoimmune diseases
* Suspected or confirmed infectious context, including virale infection VIH, VHC, VHB
* Coagulation disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-04-06 (Actual); Primary Completion 2016-01-15 (Actual); Study Completion 2016-01-15 (Actual)

PRIMARY OUTCOMES:
Measuring the expression level of markers (Gama actine, Desmine, Connexine-43, and Ocytocine receptor) by Westernblotting | up to 2 months
  Demonstrate in vitro the capacity of a Il-1B stimulus to induce the differentiation of the myometrial cells toward a hyperplasia phenotype, and that the answer depends on whether this is cells from normal weight women or obese women before conception.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Maternité du CHU de Dijon, Dijon, Bourgogne-Franche-Comté
  - Clinique Sainte Marthe, Dijon

REFERENCES:
- [Result] Barrichon M, Hadi T, Wendremaire M, Ptasinski C, Seigneuric R, Marcion G, Delignette M, Marchet J, Dumas M, Sagot P, Bardou M, Garrido C, Lirussi F. Dose-dependent biphasic leptin-induced proliferation is caused by non-specific IL-6/NF-kappaB pathway activation in human myometrial cells. Br J Pharmacol. 2015 Jun;172(12):2974-90. doi: 10.1111/bph.13100. Epub 2015 Mar 24. PMID 25653112